CLINICAL TRIAL: NCT04411511
Title: The Influence of the Covid-19 Pandemia on the Health Behaviour of Primary School Children (and Their Parents) - COVID-19, Obesity and Lifestyle in Children
Brief Title: COVID-19, Obesity and Lifestyle in Children
Acronym: COLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1330
Record Dates: First submitted 2020-05-20; First posted 2020-06-02 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Covid-19; Obesity, Childhood; Lifestyle; Lifestyle, Healthy; Overweight, Childhood; Children, Only; Family
Keywords: children; lifestyle; pandemic; covid-19; overweight; obesity; adolescents
MeSH Terms: conditions — COVID-19; Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean children: Children between 4-18 years, living in the Netherlands.
  Interventions: Other: Exposure to the Dutch measures due to the Covid-19 pandemic.
- Children with overweight or obesity: Children between 4-18 years, living in the Netherlands. Besides inclusion from the general population, childhood expertise centres will contact their patients to pay attention to this study.
  Interventions: Other: Exposure to the Dutch measures due to the Covid-19 pandemic.

INTERVENTIONS:
Other: Exposure to the Dutch measures due to the Covid-19 pandemic. — Several measures are taken in The Netherlands, due to the Covid-19 virus and pandemic. For example, closure of schools and sportclubs, and advices to stay at home as much as possible. During the pandemic, several measures also will be scaled down.

SUMMARY:
This study aims to evaluate the impact of the COVID-19 pandemic and its measures on lifestyle in Dutch children between 4 - 18 years.

DETAILED DESCRIPTION:
The threat of the severe acute respiratory syndrome coronavirus (SARS-CoV-2, from here onward mentioned as COVID-19) and the national measures to restrict transmission of COVID-19 in the Dutch population have caused a radical change in the daily life of Dutch citizens. Closing of schools and public locations, even as the public order for social distancing and self-isolation, is affecting the daily structure and lifestyle habits of Dutch children greatly. These radical changes in the current situation could yield important information regarding the health behaviour of children and their families. Knowledge of these changes and their effects on the health behaviour of these children and their families could influence future interventions and regulations regarding health behaviour. Current (preliminary) prevalence figures show that up to 80% of patients infected with COVID-19 are overweight or obese, indicating that being overweight or obese could be a potential adverse predisposition in the course of a COVID-19 infection. In the light of this (and possible future) pandemic, it is important to investigate the effects of the COVID-19 pandemic on the health behaviour i.e. lifestyle of children (aged between 4 and 18 years) and their families and especially the effects on possible weight gain during the COVID-19 pandemic. Earlier studies demonstrated that in particular children with overweight/obesity gain weight in situations when schools close such as during summer holidays and also during (economic) crisis. It is of importance to investigate the effects of the Corona-crisis in particular in these children with a high health risk.

This study aims to evaluate the impact of the COVID-19 pandemic and its measures on lifestyle in lean children and children with overweight and obesity. It evaluates differences in subgroups, e.a. lean/overweight children, socio-economic status, gender and age.

Study design is a mixed-methods study. Children and/or parents will receive online questionnaires regarding lifestyle during governemantal measures due to the Covid-19 pandemic, such as closure of schools and sportclubs.

In addition, several children and parents will be interviewed about the changes in lifestyle, and their needs for working on lifestyle, during the pandemic, for in-depth qualitative information.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 - 18 years.
* Living in The Netherlands.

Exclusion Criteria:

* No signed informed consent by relevant parties (parents of children aged below 12 years, parents and or children aged between 12 and 16 years, or children aged 16 years and older)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children (boys and girls, aged between 4 and 18 years) and their parents living in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2022-11-12 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight child | Every 2 weeks until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  Weight development of the child. Weight (in kg) will be measured using scales at home, with clear instructions.
Change in weight parents | Every 2 weeks until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs, hereafter: "coronacrisis-period"). Three months after the "measures"-period, 1 follow-up moment.
  Weight development of the parents. Weight (in kg) will be measured using scales at home, with clear instructions.

SECONDARY OUTCOMES:
Eating behaviour | Every month until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  eating behaviour during measures due to the coronacrisis, measured with an online questionnaire.
Symptoms | Every 2 weeks until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  COVID-19 related symptoms and adherence to governmental measures, measured with an online questionnaire.
Day structure | Every month until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  Daystructure of children during the coronacrisis, measured with an online questionnaire.
Physical activity | Every month until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  Physical activity behaviour children during the coronacrisis, measured with the Baecke questionnaire.
Screentime | Every month until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  Screentime during the the coronacrisis, measured with an online questionnaire.
Online possibilities | Every month until end of the Dutch governement measures affecting children (e.g. fully opening of the schools and sportclubs). Three months after the "measures"-period, 1 follow-up moment.
  Online possibilities for working on a healthy lifestyle, such as challenges regarding nutrition and physical activity, measured with an online questionnaire.
Quality of life in children | Once in first month of the study and once within three months after COVID-19 measures are scaled down.
  Quality of life during the coronacrisis, measured with the Kidscreen-27.
Parenting practices | Once in first month of the study and once within three months after COVID-19 measures are scaled down.
  Parenting practices regarding eating behaviour and physical activity, measured with a questionnaire.

OTHER OUTCOMES:
Qualitative data on lifestyle in children | Up to approximately 1 year
  Qualitative data on lifestyle in children during the coronacrisis, by semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Anita CE Vreugdenhil, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Lubrecht J, Arayess L, Reijnders D, Hesselink ML, Velde GT, Janse A, von Rosenstiel I, van Mil EGAH, Verweij M, Vreugdenhil ACE. Weight Gain in Children during the COVID-19 Pandemic and the Protective Effect of Lifestyle Intervention in Children with Obesity. Obes Facts. 2022;15(4):600-608. doi: 10.1159/000525298. Epub 2022 May 31. PMID 35640561